CLINICAL TRIAL: NCT06410560
Title: "Culture is Care: Training Workshop for Care Workers" Study
Brief Title: Culture is Care: Training Workshop for Care Workers (VerbaCurant)
Acronym: VerbaCurant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Collaborators: Compagnia di San Paolo (Other); Scuola Holden Contemporary Humanities (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ASO.IRFI.21.02
Record Dates: First submitted 2024-05-02; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Empathy; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training workshop with hands-on laboratory (Experimental): Participants will undergo a training course for a total of 12 hours: 4 FAD + 8 in the laboratory. They will receive theoretical narrative medicine education with 4 hours of distance education and a practice course of storytelling and creative writing whit 8 hours of distance education in small groups, enabling discussion and interaction among participants.
  Interventions: Other: Training about storytelling and creative writing: 12 hours
- Brief training course (Placebo Comparator): Participants will undergo a training course for a total of 4 FAD hours. They will receive theoretical narrative medicine education with 4 hours of distance education.
  Interventions: Other: Training only about theoretical narrative medicine: 4 hours

INTERVENTIONS:
Other: Training about storytelling and creative writing: 12 hours — Participants in training courses on creative writing and storytelling.
  Arms: Training workshop with hands-on laboratory
Other: Training only about theoretical narrative medicine: 4 hours — Participants in training courses on only theoretical narrative medicine.
  Arms: Brief training course

SUMMARY:
The study aims to measure the empathic capacity of healthcare professionals belonging to the Alessandria Hospital, by applying validated measuring instruments, before and after a specific training intervention. The secondary objective is to assess how the training initiative impacts on subjects with a different attitude towards cultural participation.

DETAILED DESCRIPTION:
The aim of this project is to identify how a medical humanities intervention can act on the empathic capacity of carers through culture. One of the aims is to introduce an additional element to overcome the problems about language, prejudices, legitimisation by stakeholders who do not yet recognise the value and importance of projects promoting the relationship between culture, wellbeing and health. "Verba Curant" is aimed at generating cultural value, with the hope that it can unite the different professional fields involved and become the heritage of the community.

The project of the Alessandria Hospital Centre in collaboration with the Holden School intends to launch a series of actions aimed at promoting the beneficial impact of culture, in particular storytelling, on the caregivers and patients of the Alessandria Hospital in order to measure how much cultural enjoyment can impact on health literacy. It is planned to define a methodological tool useful for making care workers aware of the importance of culture and dialogue with patients, as well as being able to measure their degree of literacy. The tool will be the object of a widespread training action on care workers, which will also involve all the stakeholders involved in the transmission of health information to patients.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals related to the Alessandria Hospital

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Empatic capacity | Before the intervention (Baseline/T0) and immediately after the intervention (Final/T1)
  Assessment of the empathic capacity of health workers through the Jefferson of Empathy scale in two groups (treated and controls).
Wellbeing | Before the intervention (Baseline/T0) and immediately after the intervention (Final/T1)
  Assessment of the wellbeing level of health workers through the PGWBI questionnaire in two groups (treated and controls).

CONTACTS AND LOCATIONS:
Overall Officials: Marinella Bertolotti, Biologist, Principal Investigator — Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo
Locations (1):
- Azienda Ospedaliera SS Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont, Italy